CLINICAL TRIAL: NCT01227512
Title: Phase 3b, Multicenter, Randomized, Single-blind, Parallel Group Trial of the Effects of Titrated Oral SAMSCA(r) (Tolvaptan) 15, 30, or 60 mg QD Compared to Placebo Plus Fluid Restriction on Length of Hospital Stay and Symptoms in Subjects Hospitalized With Dilutional Hyponatremia
Brief Title: Effects of Tolvaptan vs Fluid Restriction in Hospitalized Subjects With Dilutional Hyponatremia
Acronym: SALACIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment challenges and results of interim futility analysis, which showed less than likely to achieve primary endpoint goal-length of hospital stay.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 156-08-275
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Hyponatremia; Dilutional Hyponatremia; Inappropriate ADH Syndrome
Keywords: Hyponatremia; Dilutional Hyponatremia; Euvolemic Hyponatremia; Hypervolemic Hyponatremia; Fluid Restriction; Tolvaptan
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan 15-60mg (Experimental): Oral tablet without fluid restriction. After the initial dose, daily dose may be titrated based on response.
  Interventions: Drug: tolvaptan
- Fluid Restriction (Active Comparator): Placebo tablet with prescribed fluid restriction. After the initial dose, level of fluid restriction may titrated based response.
  Interventions: Other: Fluid Restriction

INTERVENTIONS:
Drug: tolvaptan — 15 mg titrated to 30 mg then 60 mg once daily as oral tablet for up to 7 days based on response.
  Other Names: SAMSCA; OPC-41061; OPC-156
  Arms: Tolvaptan 15-60mg
Other: Fluid Restriction — Placebo tablet once daily with prescribed daily fluid intake of 1500 mL, then intensifying to 2 lower volumes of fluid intake for up to 7 days based on response.
  Since all particpants were blinded to treatment, titration to stricter fluid restriction followed the same algorithm as tolvaptan, increasing both the level of fluid restriction and increasing the placebo "dose"
  Arms: Fluid Restriction

SUMMARY:
The purpose of this study is to determine if hospitalized patients with symptomatic hyponatremia treated with tolvaptan are in the hospital for less time than patients treated with fluid restriction. The study will also test if tolvaptan is better than fluid restriction in treating the symptoms of hyponatremia in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Hyponatremia in clinically euvolemic or hypervolemic states, defined as serum sodium < 130 mEq/L prior to randomization
* Clinically significant symptoms of hyponatremia, defined as a CGI-S score between 3-6, inclusive
* Female subjects of child bearing potential who agree to remain abstinent or to practice double-barrier forms of birth control from screening through 30 days following first dose on IMP

Exclusion Criteria:

* Women who are pregnant or breast feeding, and females of childbearing potential who are not using acceptable contraceptive methods (such as barrier contraceptives or methods that result in a failure rate of less than 1%)
* Hyponatremia in hypovolemic states, defined as the presence of clinical and historical evidence of extracellular fluid volume depletion, including but not limited to skin turgor, orthostatic changes in blood pressure or heart rate, dry mucous membranes, or a response to IV saline challenge
* Subjects who are likely to require prolonged hospitalization for reasons other than hyponatremia, eg. new femoral fracture, surgeries requiring extended recovery
* Recent prior treatment for hyponatremia: hypertonic saline (including normal saline challenge) (within 8 hours of baseline) or urea, lithium, demeclocycline, conivaptan or tolvaptan (within 4 days of baseline). Includes any treatment, other than fluid restriction for the purpose of increasing serum sodium.
* Hyponatremia symptoms of a severity (eg, CGI = 7) such that they require immediate intervention with hypertonic saline; or are expected to require such therapy within 48 hours
* Causes of neurological symptoms which are attributable to psychological (psychosis), structural (dementia of the Alzheimer's type, stroke, transient ischemic attack, multi-infarct dementia) or other metabolic causes (eg. hyper- or hypo-: oxemia, glycemia, calcemia, ammonemia, etc)
* Acute and transient hyponatremia associated with head trauma or severe neurological injury (eg. stroke, subdural hematoma)or the use of recreational drugs.
* History of hyponatremia known to be due to severe, untreated hypothyroidism/adrenal insufficiency
* Subjects with psychogenic polydipsia
* Systolic arterial blood pressure < 90 mmHg at screening
* History of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benazepril), or tolvaptan
* History of drug or medication abuse within the 3 months prior to screening, or current alcohol abuse
* Uncontrolled diabetes mellitus defined as glucose > 300 mg/dL [16.7 mmol/L]
* Current urinary tract obstruction (eg, obstructive benign prostatic hypertrophy)
* Current condition of anuria
* Serum creatinine > 3.5 mg/dL at screening
* Terminally ill or moribund condition with little chance of short-term (eg, 30 day) survival
* Subjects whose hyponatremia is the result of any medication that can safely be withdrawn (examples of drugs often not withdrawn include: anticonvulsants [eg, carbamazepine] and antipsychotics [eg, haloperidol])
* Patients receiving DDAVP within 2 days of screening
* Patients with history of active variceal bleeding within the past 30 days, without prior approval from sponsor medical monitor
* Participation in another investigational drug trial within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Dandurand, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (49):
- United States (49):
  - Otsuka Investigational Site, Birmingham, Alabama
  - Otsuka Investigational Site, Mobile, Alabama
  - Otsuka Investigational Site, Azusa, California
  - Otsuka Investigational Site, Banning, California
  - Otsuka Investigational Site, Culver City, California
  - Otsuka Investigational Site, Fountain Valley, California
  - Otsuka Investigational Site, Los Angeles, California
  - Otsuka Investigational Site, Northridge, California
  - Otuska Investigational Site, Orange, California
  - Otsuka Investigational Site, Yorba Linda, California
  - Otsuka Investigational Site, Denver, Colorado
  - Otsuka Investigational Site, Washington D.C., District of Columbia
  - Otsuka Investigational Site, Jacksonville, Florida
  - Otsuka Investigational Site, Orlando, Florida
  - Otsuka Investigational Site, Port Charlotte, Florida
  - Otsuka Investigational Site, Savannah, Georgia
  - Otsuka Investigational Site, Elizabethtown, Kentucky
  - Otsuka Investigational Site, Baltimore, Maryland
  - Otsuka Investigational Site, Springfield, Massachusetts
  - Otsuka Investigational Site, Saginaw, Michigan
  - Otsuka Investigational Site, Southfield, Michigan
  - Otsuka Investigational Site, Minneapolis, Minnesota
  - Otsuka Investigational Site, Rochester, Minnesota
  - Otsuka Investigational Site, Jackson, Mississippi
  - Otsuka Investigational Site, St Louis, Missouri
  - Otsuka Investigational Site, Grand Island, Nebraska
  - Otsuka Investigational Site, Omaha, Nebraska
  - Otsuka Investigational Site, Haddon Heights, New Jersey
  - Otsuka Investigational Site, Newark, New Jersey
  - Otsuka Investigational Site, Buffalo, New York
  - Otsuka Investigational Site, Jamaica, New York
  - Otsuka Investigational Site, New York, New York
  - Otsuka Investigational Site, The Bronx, New York
  - Otsuka Investigational Site, Cincinnati, Ohio
  - Otsuka Investigational Site, Cleveland, Ohio
  - Otsuka Investigational Site, Columbus, Ohio
  - Otsuka Investigational Site, Fairfield, Ohio
  - Otsuka Investigational Site, Toledo, Ohio
  - Otsuka Investigational Site, Oklahoma City, Oklahoma
  - Otsuka Investigational Site, Bethleham, Pennsylvania
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, West Reading, Pennsylvania
  - Otsuka Investigational Site, Providence, Rhode Island
  - Otsuka Investigational Site, Galveston, Texas
  - Otsuka Investigational Site, Houston, Texas
  - Otsuka Investigational Site, Mission, Texas
  - Otsuka Investigational Site, San Antonio, Texas
  - Otsuka Investigational Site, Fairfax, Virginia
  - Otsuka Investigational Site, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 191 participants were recruited at 81 study sites in the United States (US). A total of 124 participants were randomised to treatment.
Pre-assignment Details: Participants randomized 1:1 to tolvaptan (15 mg/day,titrated to 30 mg/day or 60 mg/day) without fluid restriction or placebo with titrated fluid restriction (500 to 1500 mL/day). Stratified based on severity of baseline symptoms (3-4, or 5-6 on the Clinical Global Impression of Severity and study center. All partipants were blinded to treatment.
Groups:
- Tolvaptan 15-60 mg/Day: Oral tablet without fluid restriction. After the initial dose, daily dose was to be titrated to 30 mg/day or 60 mg/day based on serum sodium response.
- Placebo: Placebo tablet with prescribed fluid restriction. After the initial dose, level of fluid restriction may be titrated based on serum sodium response.
Period: Overall Study
Arm/Group | Tolvaptan 15-60 mg/Day | Placebo
Started | 66 | 58
Completed | 53 | 48
Not Completed | 13 | 10
Not completed — Physician Decision | 6 | 6
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Participant met withdrawal criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan 15-60 mg/Day | Placebo | Total
Number analyzed (Participants) | 66 | 58 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (15.8) | 67.7 (15.6) | 66.7 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 37 | 24 | 61

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay (LoS)
Description: LoS was time to clinically ready to be hospital discharged (CRBD) from study treatment initiation, disregarding prolonged hospitalization due solely to social factors.
Time Frame: 45 days
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Tolvaptan 15-60mg/Day: Oral tablet without fluid restriction. After the initial dose, daily dose was to be titrated to 30 mg/day or 60 mg/day based on serum sodium response.
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 66 | 55
Days | 3.5 [3.0 to 4.5] | 4.0 [3.5 to 5.0]
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.9495, Generalized Wilcoxon Test — The alpha level was set at 0.05; Participants who used rescue therapy within first 7 days of treatment period were censored at time they started the rescue therapy

2. Secondary Outcome: Change From Baseline to 48 Hour Post Dose in Clinical Global Impression-Severity (CGI-S) of Hyponatremia Symptoms.
Description: Change from baseline in blinded rater assessed CGI-S at 48 hours post-first dose or at discharge/rescue therapy, if earlier was assessed.
  The CGI-S is a one-question rating scale which was as follows: "Considering your total clinical experience with hyponatremia symptoms in this particular population, how symptomatic is the patient at this time?" 0=not assessed; 1=normal, not at all symtpmatic; 2=borderline symptomatic; 3=mildly symptomatic; 4=moderately symptomatic; 5=markedly symptomatic; 6=severely symptomatic; 7=among the most severly symptomatic patients.
Time Frame: Baseline to 48 hours post dose
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation.
  Data were missing for one participant in the Tolvaptan group.
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Placebo: Placebo tablet with prescribed fluid restriction. After the initial dose, level of fluid restriction be may titrated based on serum sodium response.
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 65 | 55
Units on a scale
  Baseline | 4.0 [2.0 to 6.0] | 4.0 [3.0 to 6.0]
  48 hours post dose | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0]
  Change from baseline | -1.0 [-3.0 to 3.0] | -1.0 [-3.0 to 3.0]
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.1460, ANCOVA — alpha level was set at 0.05. p-value was derived from an ANCOVA model with treatment and clinical center as factors and baseline value as covariate; Includes factors of treatment, study center and covariate baseline; Mean Difference (Final Values) = -0.30, 95% CI [-0.70 to 0.11]

3. Secondary Outcome: Change From Baseline to 24 and 72 Hours Post Dose in CGI-S of Hyponatremia Symptoms.
Description: Change in CGI-S of hyponatremia symptoms from pretreatment baseline at 24 and 72 hours post-first dose, or at discharge/rescue therapy if earlier was assessed.
  The CGI-S is a one-question rating scale which was as follows: "Considering your total clinical experience with hyponatremia symptoms in this particular population, how symptomatic is the patient at this time?" 0=not assessed; 1=normal, not at all symtpmatic; 2=borderline symptomatic; 3=mildly symptomatic; 4=moderately symptomatic; 5=markedly symptomatic; 6=severely symptomatic; 7=among the most severly symptomatic patients.
Time Frame: Baseline to 24 and 72 hours post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 65 | 55
Units on a scale
  Baseline | 4.0 [2.0 to 6.0] | 4.0 [3.0 to 6.0]
  24 hours post-dose | 3.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0]
  Change from baseline at 24 hours | -1.0 [-3.0 to 3.0] | -1.0 [-3.0 to 2.0]
  72 hours post-dose | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0]
  Change from baseline at 72 hours | -2.0 [-4.0 to 3.0] | -1.0 [-4.0 to 4.0]
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; P value corresponds to 24 hours post-dose; Test type: Superiority or Other; p = 0.3150, ANCOVA; P-value was derived from an ANCOVA model with treatment and clinical center as factors and baseline value as covariate; Mean Difference (Final Values) = -0.19, 95% CI [-0.57 to 0.19]
Statistical Analysis 2: Comparison: Tolvaptan 15-60mg/Day vs Placebo; P value corresponds to 72 hours post-dose; Test type: Superiority or Other; p = 0.5381, ANCOVA; P-value was derived from an ANCOVA model with treatment and clinical center as factors and baseline value as covariate; Mean Difference (Final Values) = -0.13, 95% CI [-0.57 to 0.30]

4. Secondary Outcome: Change From Baseline to 48 Hours Post Dose in Clinical Global Impression - Improvement (CGI-I) Score of Hyponatremia Symptoms.
Description: Change in CGI-I score at 48 hours post-first dose or discharge/rescue therapy, if earlier was assessed.
  The CGI-I is a one-question rating scale where the participant is asked to rate total improvement whether or not, in their judgment, it is due entirely to trial treatment. Compared to his/her condition at admission to the trial, how much has he/she changed? 0=not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse
Time Frame: Baseline to 48 hours post dose
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation. Data were not available for 2 participants in the tolvaptan group.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 64 | 55
Units on a scale | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.2702, Cochran-Mantel-Haenszel — P-value was derived from a Cochran-Mantel-Haenszel (CMH) row mean scores test; Mean Difference (Final Values) = -0.26, 95% CI [-0.73 to 0.21]

5. Secondary Outcome: Change From Baseline in Serum Sodium Concentration (24 Hour Area Under the Curve [AUC]).
Description: Average 24 hour AUC of serum sodium concentration change from baseline, from Day 1 Hour 0 up to 72 hours post-first dose was assessed.
  A serum sodium sample was drawn at pre-treament and 8, 24, 48, and 72 hours post-first dose. Serum sodium was also assessed between 36 and 72 hours after the last dose.
  Analysis of AUC was for daily average AUC, hence the units or AUC are mEq/L/24 hours.
Time Frame: 0 to 72 hours
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation.
  Data were missing for 3 participants in the tolvaptan group and 1 participant in the placebo group.
Measure: Least Squares Mean (Full Range); unit: mEq/L
Groups:
- Placebo: Placebo tablet with prescribed fluid restriction. After the initial dose, level of fluid restriction may titrated based on serum sodium response.
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 63 | 54
mEq/L | 3.90 [-26.9 to 13.04] | 0.13 [-20.6 to 11.76]
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0019, ANCOVA — P-value was derived from an ANCOVA model with treatment and clinical center as factors and baseline value as covariate; Mean Difference (Final Values) = 3.77, 95% CI [1.43 to 6.11]

6. Secondary Outcome: Time to First 2-point Improvement in CGI-S Score.
Description: CGI-S data up to 72 hours were used to identify 2-point improvements. Please refer to outcome measure 2 for details on the scale. For the analysis of time to first 2-point improvement in CGI-S, CGI-S data up to Hour 72 were used to identify 2-point improvements. Data for participants who received rescue therapy were censored at the time of receiving rescue therapy. For participants who were discharged before Hour 72 without reaching 2-point improvement in CGI-S, data were censored at the time of discharge. Other participants who did not reach the 2-point improvement during the 72 hours also had their data censored at their last CGI-S observations within 72 hours.
Time Frame: Up to 72 hours
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation. Data were missing for 1 participant in the tolvaptan group and 3 participants in the placebo group.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 65 | 55
Hours | 51 [49 to 72] | 69 [49 to 73]
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.5128, Generalized Wilcoxon Test — p-value was derived from Generalized Wilcoxon test stratified by treatment. Participants who received rescue therapy were censored at the time of receiving rescue therapy

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression-Improvement (CGI-I) Score Improved to a Score of 1 or 2.
Description: Percentage of responders (defined as CGI-I score of 1 = very much improved or 2 = much improved) at 48 hours post-first dose, or at discharge/rescue therapy, if earlier. Participants given rescue therapy were given a score of 7.
Time Frame: 48 hours post dose
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation. Data were missing for 2 participants in the tolvaptan group and 3 participants in the placebo group.
Measure: Number; unit: Percentage of participants
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 64 | 55
Percentage of participants | 57.8 | 52.7
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.5795, Cochran-Mantel-Haenszel — P-value was derived using a CMH test stratified by hyponatremia symptoms severity; Relative Risk = 1.10, 95% CI [0.79 to 1.52]

8. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy for Hyponatremia
Description: Percentage of participants requiring rescue therapy within first 7 days of treatment for hyponatremia.
Time Frame: 7 days
Population: Analysis was performed on the modified intent-to-treat population (MITT) which included all randomized participants who received at least one dose of study drug regardless of any protocol violation. Data were missing for 3 participants in the placebo group.
Measure: Number; unit: Percentage of participants
Arm/Group | Tolvaptan 15-60mg/Day | Placebo
Number analyzed (Participants) | 66 | 55
Percentage of participants | 3.03 | 9.09
Statistical Analysis 1: Comparison: Tolvaptan 15-60mg/Day vs Placebo; Test type: Superiority or Other; p = 0.1568, Cochran-Mantel-Haenszel — p-value was derived using a CMH test stratified by hyponatremia symptoms severity; Relative Risk = 0.33, 95% CI [0.07 to 1.65]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the Informed Consent Form was signed up to 45 days after study drug administration.
Description: The same event may appear as both an adverse event (AE) and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tolvaptan 15-60 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 18/66 | 9/55
Other Adverse Events (participants affected / at risk) | 52/66 | 43/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan 15-60 mg/Day (N=66) | Placebo (N=55)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tuberculosis of central nervous system (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rapid correction of hyponatraemia (Surgical and medical procedures) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan 15-60 mg/Day (N=66) | Placebo (N=55)
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 5 | 3
Oedema peripheral (General disorders) | 4 | 4
Pyrexia (General disorders) | 3 | 3
Heart rate increased (Investigations) | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hypotension (Vascular disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No